CLINICAL TRIAL: NCT01420692
Title: The Effects of Insulin Detemir and Gliclazide-MR Treatments in Addition to Life-style Modification and Metformin Therapy on Endothelial Functions in Patients With Type 2 Diabetes : An Open-labelled Randomized Prospective Study
Brief Title: The Effects of Insulin Detemir and Gliclazide-MR Treatments on Endothelial Functions in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: Hacettepe University (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ugur Unluturk, Medical Doctor, Endocrinology and Metabolism, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110S119
Record Dates: First submitted 2010-10-28; First posted 2011-08-22 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Tip 2 DM; Endothelium; Gliclazide; Insulin detemir
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Gliclazide; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gliclazide MR (Active Comparator)
  Interventions: Drug: Gliclazide MR
- Insulin Detemir (Active Comparator): Early initiation of insulin detemir in contrast to Gliclazide MR treatment
  Interventions: Drug: Insulin Detemir

INTERVENTIONS:
Drug: Gliclazide MR — Doses between 30 mg to 120 mg/day p.o. Gliclazide MR will be arranged according to the target glycemic levels.
  Other Names: Diamicron MR
  Arms: Gliclazide MR
Drug: Insulin Detemir — Early initiation of s.c. insulin detemir in contrast to Gliclazide MR. Insulin detemir treatment will be exchanged to Gliclazide MR after 12 weeks.
  Other Names: Levemir Flexpen
  Arms: Insulin Detemir

SUMMARY:
The main purpose of this study is to analyze the effects of the addition of sulfonylurea (gliclazide MR) or ,alternatively, basal insulin (insulin detemir) to life-style modification and metformin treatment as a second step treatment in type 2 diabetes mellitus on endothelial cell functions. The second goal is to identify the effects of these treatment alternatives on body-mass index, the changes in body fat mass, insulin resistance and on the insulin secretion capacity of beta cells. The third aim of this study is to determine the success rates of these treatment alternatives on glycemic control at 6 months follow-up.

DETAILED DESCRIPTION:
The lack of enough number of randomized and controlled studies in the treatment of type 2 diabetes is the most important obstacle in recommending a single-drug or a combination treatment to the other.

The pleomorphic effects of the treatment choices other than the control of hyperglycemia in type 2 diabetes are equally important. There is yet a lack of the comparison of different treatment alternatives found in the treatment algorithms of American Diabetes Association (ADA) both in terms of the effects on hyperglycemia control as well as other pleomorphic effects. Some of these pleomorphic effects are the change in body-mass index, insulin resistance, insulin secretion capacity and the effects on endothelial functions and coagulation status.

This study is mainly prepared to analyze the effects of the addition of sulfonylurea (gliclazide MR) or alternatively basal insulin (insulin detemir) to life-style modification and metformin treatment as a second step treatment in type 2 diabetes mellitus treatment algorithm on endothelial cell functions. The second goal is to identify the effects of these treatment alternatives on body-mass index, the changes in body fat mass, insulin resistance and on the insulin secretion capacity of beta cells. The third aim of this study is to determine the success rates of these treatment alternatives on glycemic control at 6 months follow-up. This study in this sense is expected to shed the light on the decision of best treatment option as well as an essential contribution to the lacking literature in the field.

To reach these aims, 20-65 year-old patients applying to the endocrinology and the metabolism outpatient unit, having type 2 diabetes diagnoses with unregulated blood glucose levels after first step treatment (life-style modification and metformin) will be recruited and randomized either to the Gliclazide MR arm or the Insulin Detemir arm. As soon as patients in each arm reach to the target glycemic levels (0. week), basal tests showing endothelial function as well as inflammatory and coagulation status such as flow-mediated dilatation (FMD)and investigation of the peripheral blood levels of TNF-α, IL-6, MCP-1, sICAM-1, sVCAM-1, vWF, E-selectin, P-selectin, endothelin-1, PAI-1, tPA and HMW adiponectin will be performed. To investigate the insulin resistance and the changes in insulin secretory capacity of beta cells, mixed meal test will be performed and data obtained about glucose as well as insulin levels during mixed meal test will be evaluated. To identify the changes in body-fat mass, bioimpedance analyses will also be performed. All these basal tests will be repeated in each study subject, 12 weeks and 24 weeks after reaching the target glycemic levels. Patients randomized to insulin detemir arm in the beginning will only have gliclazide MR treatment after the 12.week tests are performed. The effects of continuous gliclazide MR treatment or early insulin detemir followed by gliclazide MR treatment on endothelial cell functions, inflammation and coagulation, insulin resistance, insulin secretory capacity of beta cells and body-fat mass will be evaluated by comparing the 0. week with 12. and 24. week values within each arm as well as 24. week values between arms.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic patients using at least 1000 mg/day metformin at least for 3 months
2. 7<A1C ≤ 11
3. Patients without any previous use of oral antidiabetics other than metformin or insulin
4. Between 20 to 65 years old male or female patients

Exclusion Criteria:

1. Active hepatic disease
2. Serum creatinin 1,5 mg/dl or more for males, 1,4 or more for females
3. Proliferative Diabetic Retinopathy
4. Coronary Artery Disease
5. Patients with any kind of diagnosed malignancy
6. Pregnancy and Lactation
7. Fasting C-peptide levels lower than 2.0 ng/ml
8. Smoking or drug abuse

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The evaluation of the changes in Flow-Mediated Dilatation (FMD) at 12th and 24th weeks compared to the baseline level, as a Measure of Endothelial Function | The basal, 12th and 24th week after reaching the target glycemic levels
  As soon as type 2 DM patients which were randomly recruited either to the Gliclazide MR arm or the Insulin Detemir arm reach to target glycemic levels (0. week), flow-mediated dilatation test, which is a basal tests showing endothelial function will be performed. This basal test will be reapeated in each study subject, 12 weeks and 24 weeks after reaching the target glycemic levels.
The Changes in the Peripheral Blood Levels of TNF-α, IL-6, MCP-1, sICAM-1, sVCAM-1, vWF, E-selectin, P-selectin, Endothelin-1, PAI-1, tPA and HMW Adiponectin at 12th and 24th weeks compared to the baseline level, as Measures of Inflam. and Coagulation | The basal, 12th and 24th week after reaching the target glycemic levels
  As soon as type 2 DM patients which were randomly recruited either to the Gliclazide MR arm or the Insulin Detemir arm reach to target glycemic levels (0. week), basal tests showing endothelial function as well as inflammatory and coagulation status such as flow-mediated dilatation and peripheral blood TNF-α, IL-6, MCP-1, sICAM-1, sVCAM-1, vWF, E-selectin, P-selectin, endothelin-1, PAI-1, tPA and HMW adiponectin levels will be performed. These basal tests will be reapeated in each study subject, 12 weeks and 24 weeks after reaching the target glycemic levels.

SECONDARY OUTCOMES:
Calculation of Body-mass Index, Body Fat Mass, Level of Insulin Resistance and the Insulin Secretion Capacity of Pancreatic Beta Islet Cells as Measures to Identify the Effects of Gliclazide and Insulin Detemir Treatments on Diabetes Progression | The basal, 12th and 24th week after reaching the target glycemic levels
  As soon as type 2 DM patients which were randomly recruited either to the Gliclazide MR arm or the Insulin Detemir arm reach to target glycemic levels (0. week), mixed-meal test and body-fat mass determination using bioimpedence analysis will be performed. These tests will be reapeated in each study subject, 12 weeks and 24 weeks after reaching the target glycemic levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ugur Unluturk, MD, Principal Investigator — Ankara University Medical Faculty Dept. of Endocrinology and Metabolism; Altug S Kesikli, MD. PhD., Principal Investigator — Hacettepe University Instute of Oncology Dept. of Basic Oncology
Locations (1):
- Ankara University Medical Faculty Dept. of Endocrinology and Metabolism, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: Hacettepe University Web Page — http://www.hacettepe.edu.tr/english/